CLINICAL TRIAL: NCT07360444
Title: Safety and Efficacy of Radiofrequency Ablation of Rammii Communicans Versus Annuloplasty or Both Together in Discogenic Back Pain Patients Double-Blinded Randomized Controlled Trial
Brief Title: Radiofrequency Ablation of Rammii Communicans Versus Annuloplasty in Discogenic Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esraa Fathy Radwan Abd Elzaher (Other)
Responsible Party: Sponsor-Investigator, Esraa Fathy Radwan Abd Elzaher, dr, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: rammii radiofrequency ablation
Record Dates: First submitted 2026-01-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Discogenic Back Pain Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Active Comparator): Rammii Communicans Radiofrequency Ablation
  Interventions: Procedure: radiofrequency ablation of Rammii Communicans
- group 2 (Active Comparator): Annuloplasty Radiofrequency Ablation
  Interventions: Procedure: Annuloplasty Radiofrequency Ablation
- group 3 (Active Comparator): both techniques
  Interventions: Procedure: radiofrequency ablation of Rammii Communicans; Procedure: Annuloplasty Radiofrequency Ablation

INTERVENTIONS:
Procedure: radiofrequency ablation of Rammii Communicans — Standard ASA monitoring, Fluoroscopy Sterile prep and drape Apply local anesthesia to the skin before any needle larger than 25G The coaxial view is always used to advance the needle CPR equipment and medications available 18-20G, 3.5 inch (90 mm) - 6 inch (150 mm), 5-10 mm active tip, blunt or sharp, curved radiofrequency cannula for radiofrequency ablation (RFA) Nonionic contrast Local anesthetic: 1-2 ml 1% lidocaine or 0.5% bupivacaine
  Fluoroscopy Technique, Target Localization Patient prone, Anteroposterior (AP) image Square off vertebral endplates Turn the C-arm obliquely toward the ipsilateral side, approximately 30°, until the transverse process overlaps the lateral margin of the vertebral body (Fig. 5.2a-c). Entry point is just below the transverse process, in line with the lateral edge of the vertebral body, about 6-7 cm off midline, depending on body habitus Needle entry at lumbar level chosen Coaxial view until bony contact is made with the vertebral body Lateral v
  Arms: group 1; group 3
Procedure: Annuloplasty Radiofrequency Ablation — Standard ASA monitoring, Fluoroscopy Sterile prep and drape Apply local anesthesia to the skin before any needle larger than 25G The coaxial view is always used to advance the needle CPR equipment and medications available 18-20G, 3.5 inch (90 mm) - 6 inch (150 mm), 5-10 mm active tip, blunt or sharp, curved radiofrequency cannula for radiofrequency ablation (RFA) Nonionic contrast Local anesthetic: 1-2 ml 1% lidocaine or 0.5% bupivacaine Patient prone, Anteroposterior (AP) image Square off the vertebral endplates Turn the C-arm obliquely toward the ipsilateral side, approximately (20-30°), until the SAP (superior articular process) of the lower vertebra in the middle of the vertebral body Needle entry at lumbar level chosen Coaxial view until bony contact is made with the SAP of the vertebral body Once touched, SAP "wiggle" laterally, constantly keeping the needle contacting the SAP with fluoroscopy control to the target location In the Lateral view, the tip of the needle is at th
  Arms: group 2; group 3

SUMMARY:
Aim of the study

Comparing the safety, efficacy, pain reduction, and functional disability between Ramii communicans radiofrequency versus Annuloplasty versus combined both techniques in patients with discogenic low back pain

Patient and methods

• Study design: Prospective, randomized, double-blinded control clinical trial study.

• Study suite: The study will be conducted in the pain management unit at the Department of Anesthesia and Pain Management, Assiut University Hospital, after approval of the local ethical committee.

• Time of study: from January 2026 till the recruitment of all patients.

The PICOT algorithm is preliminarily pointed out:

* P (Population): patients complaining of Discogenic back pain with failed conservative treatment
* I (Intervention) Patients scheduled for Rammii Communicans Radiofrequency Ablation
* C (Comparison): patients scheduled for Annuloplasty Radiofrequency Ablation
* O (Outcomes): Assess safety, Efficacy, pain reduction (assessed by Numeric Rating Scale), functional disability (assessed by Oswestry Disability Index), and Depression score (SF-36) between the two groups
* T (Timing): 2weeks,1 month,3 months, and 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 18 years or older
* Chronic LBP persisted for more than three months
* Failed medical treatment
* Axial LBP with or without leg radicular pain experienced pain exacerbation by sitting (intolerance to sitting), bending forward, coughing or sneezing, and partially relieved with lateral recumbent position, standing, or walking.
* Patients with a Numeric Rating Scale of pain severity of five points or higher, specifically to the daily LBP, were included in the study.
* The examination criteria for the study included tenderness on deep pressure of the spine process at the level of the degenerated disc and no neurological motor deficits.
* The magnetic resonance imaging (MRI) criteria required images to show clear evidence of degenerative disc disease in one or two-disc levels that include a high intensity zone (HIZ) in the posterior annulus and dark disc with or without loss of height

Exclusion Criteria:

* Encompassed patients with clinical evidence of progressive motor neurological deficits,
* MRI evidence of intervertebral disc herniation measuring 4 mm or more, sequestration, extrusion, disc space collapse, or spondylolisthesis at the symptomatic level.
* Patients with moderate to-severe central spinal canal or foraminal stenosis,
* Previous lumbar surgery at the same treatment level,
* Spinal fractures, deformities
* Infections or tumors
* Patients with psychotic illnesses, uncontrolled diabetes, advanced hepatic conditions, current pregnancy, recent delivery (within three months of consent), intent to become pregnant during the study period, and local sepsis or skin inflammation in the back region.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients who were 18 years or older
Enrollment: 90 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain Intensity Changes | 2 weeks,1 month, 3 months, and 6 months.
  Change from baseline in the Numeric Rating Scale (NRS; 0-10) A Numeric Rating Scale (NRS) is a simple, widely used tool (often 0-10) for quantifying subjective experiences like pain or satisfaction, where 0 means none/worst and 10 means worst/best, allowing for easy tracking of changes, especially in healthcare for assessing pain intensity, treatment response, and function over time. It's used in research and clinical settings to get a numerical measure of abstract feelings, with anchors like "no pain" (0) and "worst imaginable pain" (10)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kallewaard JW, Terheggen MA, Groen GJ, Sluijter ME, Derby R, Kapural L, Mekhail N, van Kleef M. 15. Discogenic low back pain. Pain Pract. 2010 Nov-Dec;10(6):560-79. doi: 10.1111/j.1533-2500.2010.00408.x. Epub 2010 Sep 6. PMID 20825564
- [Result] Oh WS, Shim JC. A randomized controlled trial of radiofrequency denervation of the ramus communicans nerve for chronic discogenic low back pain. Clin J Pain. 2004 Jan-Feb;20(1):55-60. doi: 10.1097/00002508-200401000-00011. PMID 14668658